CLINICAL TRIAL: NCT01617044
Title: Probiotics in the Treatment of Iron Deficiency in Children With Restless Leg Syndrome-A Double-blind, Randomized Controlled Study
Brief Title: Probiotics in the Treatment of Iron Deficiency in Children With Restless Leg Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Probiotics_Iron Defieciency
Record Dates: First submitted 2012-03-08; First posted 2012-06-12 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Iron Deficiency; Restless Leg Syndrome
Keywords: Iron; Deficiency; Restless; Leg
MeSH Terms: conditions — Iron Deficiencies; Restless Legs Syndrome; Psychomotor Agitation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 1. iron 3 mg/kg/day elemental iron FeSO4 up to 45 mg (dose to be determined by PI)
  2. + vitamin C-250 mg chewable tab
  3. + probiotics lactobacillus plantarum 299 (1x10x8 colony forming units)
  Interventions: Dietary Supplement: Probiotics
- Control (Placebo Comparator): 1. iron 3 mg/kg/day elemental iron FeSO4 to 45 mg
  2. + vitamin C-250 mg chewable tab
  3. + placebo (identical capsule)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — probiotics lactobacillus plantarum 299 (1x10x8 colony forming units)
  Arms: Treatment
Dietary Supplement: Placebo — Placebo
  Arms: Control

SUMMARY:
A double-blind randomized controlled trial comparing iron plus vitamin C plus probiotic (lactobacillus plantarum 299) to iron plus vitamin C plus placebo in correcting the iron deficiency in children with Restless leg syndrome (RLS) and iron deficiency. One hundred children with diagnosis of RLS will be recruited over a two- year period.

DETAILED DESCRIPTION:
Project Summary:

Iron deficiency is the most common micronutrient deficiency in the world and is associated with significant adverse health effects including: cognitive deficits, immune deficiency, anemia, fatigue, and increased mortality. RLS affects 5 to 10% of adults in the United States and 2% of children. The prevalence of RLS in children with attention deficit hyperactivity disorder (ADHD) is estimated to be 12 to 35%. Iron deficiency has been recognized as an important factor in RLS, and the current recommendation for adults and children with RLS is to maintain serum ferritin level above 50 mcg/l. A common problem in the treatment of iron deficiency is that oral iron is poorly absorbed.

Probiotics are a group of microorganisms that benefit the host and are available naturally in fermented foods or as oral supplements. Naturally occurring probiotics, such as yogurt have been used to promote human health for millennia. Probiotic oral supplements have been proven effective and are currently approved for use in pediatrics in the treatment of: acute diarrhea, antibiotic associated diarrhea, and atopy associated with cow milk allergy; and there is some evidence that probiotics may be useful in the treatment of irritable bowel syndrome and necrotizing enterocolitis. In studies in adults, and in cell culture experiments, probiotics have improved iron absorption, but this question has never been studied in children.

Relevance:

This study proposes to compare the standard treatment for iron deficiency in children (supplemental iron plus vitamin C) with RLS; to supplemental iron plus vitamin C plus probiotics in a randomized, double-blind randomized controlled trial.

Specific Aims:

1. To improve the treatment of iron deficiency using oral iron, vitamin C, and probiotics in children with RLS and iron deficiency.
2. To evaluate the safety and monitor for adverse side effects during treatment with probiotics in children with RLS and iron deficiency.

Research Question:

The research question that this study will address is whether the addition of a specific strain of probiotics (lactobacillus plantarum 299) to the standard treatment of iron deficiency (supplemental iron + Vitamin C) will improve the treatment of iron deficiency. Children with RLS are the study population because RLS is a common diagnosis seen in our sleep center, iron deficiency is a known trigger for RLS, and the current standard of care in the evaluation of patients with RLS is to check serum ferritin level at the time of diagnosis and to treat with supplemental iron if the serum ferritin is < 50 mcg/l. However, the implications of this study go far beyond the treatment of children with RLS and iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-18 years
* RLS defined by NIH criteria -definite or probable (see appendix)
* Serum ferritin level less than 50 mcg/l
* CRP less than 10 mg/l

Exclusion Criteria:

* Immune compromised
* Milk intolerant/allergic
* Known allergy or intolerance to probiotics for iron
* History of hematochromatosis
* IV catheter or indwelling medical device
* Chronic gastroenteritis or malabsorption

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Ferritin and CRP Levels | Collection at Baseline and at 6-weeks

SECONDARY OUTCOMES:
Restless Leg Questionnaire | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Rosen, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Rosen GM, Morrissette S, Larson A, Stading P, Griffin KH, Barnes TL. Use of a Probiotic to Enhance Iron Absorption in a Randomized Trial of Pediatric Patients Presenting with Iron Deficiency. J Pediatr. 2019 Apr;207:192-197.e1. doi: 10.1016/j.jpeds.2018.12.026. Epub 2019 Feb 4. PMID 30732996